CLINICAL TRIAL: NCT05270317
Title: Bone Graft Cultivation by Periosteal Elevation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordanian Royal Medical Services (Other)
Collaborators: The Ministry of Higher Education and Scientific Research, Jordan (Unknown)
Responsible Party: Principal Investigator, Feras Ahmed Al Ibrahim, Pediatric Orthopedic Surgeon, Jordanian Royal Medical Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPH/1/04/2020
Record Dates: First submitted 2021-12-30; First posted 2022-03-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Periosteal Elevation
Keywords: Bone graft; Periosteal Elevation; Cultivation

STUDY DESIGN:
Intervention Model Description: The study will be conducted on 18 skeletally immature patients who are suffering Bone loss problems either posttraumatic, post-tumor resection or post-infection that requires bone grafting, attending the Pediatric orthopedic Surgery Department in king Hussein Medical center.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early-Stage Group (Active Comparator): 6 patients will be allocated randomly to participate in the clinical trial with cultivation duration of 6 weeks
  Interventions: Procedure: Bone Graft Cultivation and Harvesting
- Medium -Stage Group (Active Comparator): 6 patients will be allocated randomly to participate in the clinical trial with cultivation duration of 8 weeks
  Interventions: Procedure: Bone Graft Cultivation and Harvesting
- Late -Stage Group (Active Comparator): 6 patients will be allocated randomly to participate in the clinical trial with cultivation duration of 10 weeks
  Interventions: Procedure: Bone Graft Cultivation and Harvesting

INTERVENTIONS:
Procedure: Bone Graft Cultivation and Harvesting — Participants will be randomly assigned preoperatively into three surgical groups depending on cultivation time: early-stage group, medium-stage group and late-stage group . Bone Graft Cultivation is a two-stage procedure aiming at generating new bone tissue for grafting by periosteal elevation . The first stage is the insertion of space-occupying implant which is responsible for keeping periosteal elevation for a defined time to stimulate new bone formation. The second stage is the extraction of woven bone that has been formed together with the implant.

SUMMARY:
Bone Graft Cultivation is a two-stage procedure aiming at generating new bone tissue for grafting by periosteal elevation . The first stage is the insertion of space-occupying implant which is responsible for keeping periosteal elevation for a defined time to stimulate new bone formation. The second stage is the extraction of woven bone that has been formed together with the implant. A sufficient amount of biologically highly valuable woven bone may be produced and harvested for bone grafting using periosteal elevation method. The concept of using periosteal elevation to cultivate bone has never mentioned in orthopedic literature.

Thus, this study aims to present an original experimental Interventional (Clinical Trial) on 18 skeletally immature patients. The purpose of this non-comparative study is to test, for the first time, possibility of generating bone tissue from iliac bone and to test the bioactivity of this new "Bone Graft Material" in fillings of losses of osseous substance from various origins, such as traumatic, infection, and benign tumoral causes.

Study protocol: Participants will be randomly assigned preoperatively into three surgical groups depending on cultivation time: early-stage group, medium-stage group and late-stage group . The newly bone formed bone will undergo tissue processing, and then, bone volume/tissue volume ratio, osteoid volume/tissue volume ratio, and osteocyte count per high-power field will be analyzed. In addition to histological examination, micro-CT scanning and osteoinductive factors ( bone morphogenic protein (BMP2), Fibroblast growth factor-2(FGF2), Transforming Growth Factor(TGFB1), and Insulin-like growth factor(IGF1)) assessment will be done as well

DETAILED DESCRIPTION:
Most of the current strategies for bone grafting exhibit relatively unsatisfactory results and most of them are associated with drawbacks and limitations to their use and availability, and even controversial reports about their efficacy and cost-effectiveness. Furthermore, at present there are no heterologous or synthetic bone substitutes available that have superior or even the same biological or mechanical properties compared with autogenous bone graft. Therefore, there is a necessity to develop a new treatments as alternatives or adjuncts to the standard methods used for bone grafting, in an effort to overcome these limitations, which has been a goal for many decades. autogenic bone graft is widely regarded as an ideal and the best construct for grafting procedures, autogenic bone supply osteoinductive growth factors, osteogenic cells, and a structural scaffold in most cases when used to fill bone defect or treating nonunion or other indications. However, site morbidity and constraints on obtaining large quantities limit its use. in treating large bone defects resulted from bone tumors or after resection of infected bone or dead bone after trauma raise the big need for large quantity of bone graft which is most of the times difficult to take it from the patient own reservoir. so limited amount of autologous bone graft available in such cases with the superiority of the quality of autologous bone graft. Allograft on the other hand is the next best alternative; however, immunogenic rejection with the risk of disease transmission are unresolved issues. despite that ,the synthetic bone graft materials eliminate these risks, synthetic bone grafts do not transfer osteoinductive or osteogenic elements to the host site. So ,large bone defects remain a clinical challenge in autograft or allograft transplantation. using this new method of bone cultivation would like to harvest large amounts of autologous bone graft with all advantages of osteoinductive and osteogenic cells that can solve the clinical challenge in large bone defects with minimal site morbidity.

Our understanding of bone grafting at the cellular and molecular level has advanced enormously, and is still ongoing. New methods for studying this process, such as quantitative three-dimensional microcomputed tomography analyses, finite element modelling, and nanotechnology have been developed to further evaluate the mechanical properties of bone graft at the microscopic level. In addition, advances made in cellular and molecular biology have allowed detailed histological analyses, in vitro and in vivo characterization of bone-forming cells, identification of transcriptional and translational profiles of the genes and proteins involved in the process of bone grafting and fracture repair, and development of transgenic animals to explore the role of a number of genes expressed during bone repair, and their temporal and tissue-specific expression patterns . With the ongoing research in all related fields, novel therapies have been used as adjuncts or alternatives to traditional bone-grafting methods. Nevertheless, the basic concept for managing all clinical situations requiring bone grafting, particularly the complex and recalcitrant cases, remains the same, and must be applied. Treatment strategies should aim to address all (or those that require enhancement) prerequisites for optimal bone healing, including osteoconductive matrices, osteoinductive factors, osteogenic cells and mechanical stability, following the 'diamond concept' suggested for fracture healing.

The idea of using periosteal elevation to induce bone growth and cultivate new bone for grafting came after investigators noticed that a large amount of bone grows around the K-wires that investigators use to fix the iliac bone in pelvis osteotomies in the pediatric population. In fact investigators have done thousands of pelvic osteotomies( Salter Osteotomy) over the last two decades at investigators institution in royal medical services. During pelvis osteotomy, investigators elevate the periosteum and after performing the osteotomy investigators use K-wires to fix it. Usually, these K-wires are removed after the osteotomy heals by another operation. investigators always noticed that the width of the iliac bone was 3 to 4 times the original width for the same age which means that periosteal stripping can produce more bone under the periosteal tissue and the cause of change in the bone size. This raises the idea that if investigators elevate the periosteum intentionally and create a space under it by keeping it elevated using space occupying implant, the bone will grow into that space and fill it. In theory, investigators can grow new bone into that subperiosteal space. Indeed, investigators have started to test this concept and investigators have performed Bone Cultivation using a periosteal elevation technique on five patients after taking their consent who presented to us with large long bone defects and very difficult clinical scenarios that could not heal without very good quality and quantity of bone graft material.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with Bone loss pathologies.
* Males and females between one year and 14 years.
* post-traumatic, bone cysts or tumoral cases or post-infection and congenital pseudoarthrosis that requires bone grafting

Exclusion Criteria:

* Patients with systemic illness as cardiac diseases, or mental disorders or neuromuscular disorders & hepatic patients (generally debilitating diseases).

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2021-12-19 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of new bone | 6-10 weeks
  ability to generate new bone

SECONDARY OUTCOMES:
Assessment of Qualitative Feature of the newly formed bone | 6 weeks, 8 weeks , 10 weeks
  The new bone will be assessed by micro CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Feras AL Ibrahim, MD, Principal Investigator — Royal Medical Services
Locations (1):
- Royal Medical Services, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No